CLINICAL TRIAL: NCT03319615
Title: Biological and Psychological Mediators of the Relationships Between Fat Mass, Fat-free Mass and Energy Intake
Brief Title: The Effect of Fat Mass, Fat-free Mass and Resting Metabolic Rate on Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Dr Graham Finlayson, Associate Professor, University of Leeds
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FSNHop001
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Appetitive Behavior
Keywords: Appetite; Energy Intake; Body Composition; Energy Expenditure
MeSH Terms: conditions — Appetitive Behavior

STUDY DESIGN:
Intervention Model Description: The baseline non-intervention control arm only used in the present secondary data analysis
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Habitual dietary intake (No Intervention): Habitual dietary intake
- Energy Restriction (Experimental): Match period (to comparator) of dietary energy restriction
  Interventions: Behavioral: Dietary energy restriction

INTERVENTIONS:
Behavioral: Dietary energy restriction
  Arms: Energy Restriction

SUMMARY:
The present study was based on secondary analysis using the non-intervention control conditions of five separate studies with common measures. The current analysis examine the indirect and direct effects of fat-free mass, fat mass and resting metabolic rate on energy intake in individuals at or close to energy balance.

DETAILED DESCRIPTION:
The current analysis examine the indirect and direct effects of fat-free mass, fat mass and resting metabolic rate on energy intake in individuals at or close to energy balance.

The present study was based on secondary analysis using the non-intervention control conditions of five separate studies conducted between the dates of 1998 and 2007. In total, 242 subjects (114 males; 128 females; mean body mass index = 25.6 ± 5.0 kg/m2) were included. In these studies, body composition (air displacement plethysmography), energy expenditure (indirect calorimetry and flex heart rate) and energy intake (weighed dietary records) were measured using common procedures.

ELIGIBILITY:
Inclusion Criteria:

* Weight stable (weight change of <2 kg in the previous three months)
* Non smoker
* Not dieting,
* No history of eating disorders,
* Free from disease

Exclusion Criteria:

* Taking medication known to effect metabolism or appetite
* Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 1998-01-01 (Actual); Primary Completion 2007-01-01 (Actual); Study Completion 2007-01-01 (Actual)

PRIMARY OUTCOMES:
Energy Intake- weighed dietary record method | Baseline
  Cross-sectional measurement of energy intake taken at baseline using the weighed dietary record method

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No